CLINICAL TRIAL: NCT00303641
Title: A Prospective Randomized Study of the Safety and Effectiveness of the Medtronic Resting Heart System
Brief Title: Safety and Effectiveness of the Medtronic Resting Heart Bypass System in Heart Surgery Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-04-424
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Bypass Surgery; Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass; Inflammatory reaction
MeSH Terms: conditions — Inflammation

INTERVENTIONS:
Device: Medtronic Resting Heart Bypass System

SUMMARY:
The purpose of this study is to determine if the Medtronic Resting Heart Bypass system is safer and results in less inflammatory reaction than traditional bypass machines used in coronary artery bypass surgery. We hypothesize that the new Medtronic Resting Heart System is safer and results in much less systemic inflammatory reaction in comparison to the standard cardiopulmonary bypass systems currently in use.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) has played an extremely crucial role in coronary artery bypass grafting (CABG) surgery for the past five decades. During CABG, the CPB machine enables the surgeon to stop the heart and perform the surgery in a bloodless operating field. The CPB machine essentially takes over the job of the heart by oxygenating the blood and then perfusing the entire body. In patients undergoing CABG surgery with CPB, a systemic inflammatory reaction occurs when the blood is taken out of the body and circulated through the CPB machine. This inflammatory reaction is believed to increase postoperative morbidity and prolong hospital stay. The systemic inflammatory reaction results in activation of the complement, coagulation, fibrinolytic and kallikrein cascades, it activates leukocytes and endothelial cells causing expression of adhesion molecules and results in the release of inflammatory mediators such as cytokines. This inflammatory reaction during CPB leads to vasodilation, increased interstitial fluid and can affect organs such as the heart, lungs, brain and kidneys resulting in their dysfunction(s). Elimination of CPB in patients undergoing CABG surgery has resulted in reduction of this inflammatory response. Unfortunately, not all patients are able to undergo CABG without the use of CPB.

Most conventional CPB systems also use cardiotomy suction which returns all the blood collected in the operative field back to the CPB reservoir and then eventually returns it to the patient. This blood is rich in inflammatory mediators and small particles because it has been activated by surgical trauma and by the proteins lining the wound cavity. Returning this blood back into the CPB circuit results in further circulation of inflammatory mediators. Removal of the cardiotomy suction from the CPB system could potentially decrease the inflammatory mediators and reduce the inflammatory response during CPB.

Recently, there have been attempts to decrease the inflammatory reaction caused by the use of CPB by developing better, more effective systems. The Medtronic Resting Heart System is very similar to conventional CPB systems and has been approved for clinical use both in Canada and the United States. It has some potential advantages over traditional bypass machines which include; 1)a fully closed-to-air system that does not allow an air-blood interface which could prevent blood activation, 2)it does not have cardiotomy suction and therefore prevents air, lipids or particulate emboli from being re-introduced into the patient's circulation, 3)it minimizes hemodilution by using smaller and low-prime circuits, possibly decreasing the need for postoperative blood transfusion, 4)the CPB circuit, which is the blood-contacting surface, is coated with Carmeda Bioactive Surface (a heparin bioactive surface), that mimics critical characteristics of vascular endothelium and may prevent further blood activation, and 5)it has an active venous air detector and removal device (VARD) that detects venous air and automatically removes the air which may prevent blood activation. All of these elements are potential benefits which may further reduce the morbidity and inflammation associated with CABG surgery.

Thus far to our knowledge, there have been no studies looking at the inflammatory reaction and morbidity in patients undergoing CABG procedures using more improved cardiopulmonary bypass machines. We are therefore proposing a prospective, randomized trial of the safety and effectiveness of the Medtronic Resting Heart system in CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients undergoing elective surgical coronary artery bypass grafting (CABG) with use of the cardiopulmonary bypass machine

Exclusion Criteria:

* Patients unable to provide written informed consent
* Emergency CABG surgery
* Concomitant CABG + Valvular surgery
* Off-pump CABG surgery

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-11 (Actual); Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
C-reactive protein
Cell count
Cytokine levels
Complement

SECONDARY OUTCOMES:
Postoperative blood loss, units of blood transfused, re-operation for bleeding, chest tube drainage, length of ICU stay, neurologic and renal function, infection, atrial fibrillation and overall length of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, FRCSC, Principal Investigator — Department of Cardiac Surgery, University of Western Ontario and the London Health Sciences Centre, University Hospital
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Kirklin JK, Westaby S, Blackstone EH, Kirklin JW, Chenoweth DE, Pacifico AD. Complement and the damaging effects of cardiopulmonary bypass. J Thorac Cardiovasc Surg. 1983 Dec;86(6):845-57. PMID 6606084
- [Background] Wehlin L, Vedin J, Vaage J, Lundahl J. Activation of complement and leukocyte receptors during on- and off pump coronary artery bypass surgery. Eur J Cardiothorac Surg. 2004 Jan;25(1):35-42. doi: 10.1016/s1010-7940(03)00652-3. PMID 14690730
- [Background] Edmunds LH Jr. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 1998 Nov;66(5 Suppl):S12-6; discussion S25-8. doi: 10.1016/s0003-4975(98)00967-9. PMID 9869435
- [Background] Matata BM, Sosnowski AW, Galinanes M. Off-pump bypass graft operation significantly reduces oxidative stress and inflammation. Ann Thorac Surg. 2000 Mar;69(3):785-91. doi: 10.1016/s0003-4975(99)01420-4. PMID 10750762
- [Background] Gu YJ, Mariani MA, van Oeveren W, Grandjean JG, Boonstra PW. Reduction of the inflammatory response in patients undergoing minimally invasive coronary artery bypass grafting. Ann Thorac Surg. 1998 Feb;65(2):420-4. doi: 10.1016/s0003-4975(97)01127-2. PMID 9485239
- [Background] Fransen E, Maessen J, Dentener M, Senden N, Geskes G, Buurman W. Systemic inflammation present in patients undergoing CABG without extracorporeal circulation. Chest. 1998 May;113(5):1290-5. doi: 10.1378/chest.113.5.1290. PMID 9596308
- [Background] Jewell AE, Akowuah EF, Suvarna SK, Braidley P, Hopkinson D, Cooper G. A prospective randomised comparison of cardiotomy suction and cell saver for recycling shed blood during cardiac surgery. Eur J Cardiothorac Surg. 2003 Apr;23(4):633-6. doi: 10.1016/s1010-7940(02)00834-5. PMID 12694789
- [Background] Aldea GS, Soltow LO, Chandler WL, Triggs CM, Vocelka CR, Crockett GI, Shin YT, Curtis WE, Verrier ED. Limitation of thrombin generation, platelet activation, and inflammation by elimination of cardiotomy suction in patients undergoing coronary artery bypass grafting treated with heparin-bonded circuits. J Thorac Cardiovasc Surg. 2002 Apr;123(4):742-55. doi: 10.1067/mtc.2002.120347. PMID 11986603
- [Background] Kaza AK, Cope JT, Fiser SM, Long SM, Kern JA, Kron IL, Tribble CG. Elimination of fat microemboli during cardiopulmonary bypass. Ann Thorac Surg. 2003 Feb;75(2):555-9; discussion 559. doi: 10.1016/s0003-4975(02)04540-x. PMID 12607672
- See also: London Health Sciences Centre, University Hospital, Division of Cardiac Surgery — http://www.lhsc.on.ca/cardiac_surgery